CLINICAL TRIAL: NCT03605446
Title: Protein for Life: Towards a Focused Dietary Framework for Healthy Ageing. Consumer Assessment of High Protein Biscuits
Acronym: Protein4Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newcastle University (Other)
Collaborators: University of Aberdeen (Other); University of Bristol (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Anthony Watson, Senior Research Associate, Newcastle University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 809
Record Dates: First submitted 2018-06-26; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Acceptance, Social

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind white label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Animal 12% (Experimental): Animal based protein biscuit containing 12% of total energy as protein
  Interventions: Dietary Supplement: Biscuit acceptance
- Animal 20% (Experimental): Animal based protein biscuit containing 20% of total energy as protein
  Interventions: Dietary Supplement: Biscuit acceptance
- Plant 12% (Experimental): Plant based protein biscuit containing 12% of total energy as protein
  Interventions: Dietary Supplement: Biscuit acceptance
- Plant 20% (Experimental): Plant based protein biscuit containing 20% of total energy as protein
  Interventions: Dietary Supplement: Biscuit acceptance
- Wheat biscuit (Placebo Comparator)
  Interventions: Dietary Supplement: Biscuit acceptance

INTERVENTIONS:
Dietary Supplement: Biscuit acceptance — Acceptance of high protein biscuits

SUMMARY:
As part of the Protein for Life project, design rules have been established which outline the processes which need to be considered when designing higher protein products. These design rules have been used to create a range of exemplar higher protein biscuits. Consumer feedback is needed to validate the set of design rules. This project will assess the consumer acceptance of higher protein biscuits made from plant and animal based proteins.

DETAILED DESCRIPTION:
The Protein for Life project was funded by the Research Councils UK 'Priming Food Partnerships' initiative which is supported by four councils: Biotechnology and Biological Sciences Research Council (BBSRC), Medical Research Council (MRC), Engineering and Physical Sciences Research Council (EPSRC) and Economic and Social Research Council (ESRC). The initiative supports pre-competitive research, with the aim of stimulating innovative research and technological advances of relevance to the food industry. The project has five key objectives related to the development and dissemination of guidelines for the formulation of palatable, cost effective, higher-protein foods for an ageing population.

The population of the UK is aging, and it is estimated that by 2039 more than 43% of adults will be aged over 60 (ONS 2015). One significant healthcare challenge associated with aging is sarcopenia. This refers to the decline of skeletal muscle tissue with age (Walston, 2012), and can affect physical functioning and quality of life. One reason older adults may lose muscle more easily is due to a decrease in protein intake. The current recommended daily intake of protein in the UK is 0.8g/kg body weight. However, this is an estimate for the entire population, tends to be based on a few younger individuals to determine this (Phillips, Chevalier, & Leidy, 2016). Studies which have used older adults to estimate protein and amino acid requirements have suggested that protein requirements in an older population may be well above the recommended daily intake (Rafii et al., 2015; Tang et al., 2014). Despite this, older adults do not consume increased amounts of protein. The purpose of this experiment is to explore the psychological mechanisms underlying the reduced intake of protein in older populations.

As part of the Protein for Life project, design rules have been established which outline the processes which need to be considered when designing higher protein products. These design rules have been used to create a range of exemplar higher protein biscuits. Consumer feedback is needed to validate the set of design rules. This project will assess the consumer acceptance of higher protein biscuits made from plant and animal based proteins.

As set of design rules have been established which outline the processes which need to be considered when designing higher protein products. These design rules have been used to create a range of exemplar higher protein biscuits. Consumer feedback is needed to validate the set of design rules.

Study Objective

The project will assess the consumer acceptance of 5 biscuits, each with differing protein quantities and sources. The aim is to test the design rules created in the protein for life project. Outcomes of the consumer testing will inform the project of the optimal protein source (plant or animal) and quantity for consumer acceptance.

The purpose of the trial is to assess the organoleptic properties of 4 ready to eat higher protein biscuits and one control in a healthy adult population aged 40+ years.

Methods

5 products have been developed by Campden BRI Ltd. Products have been created in a food safe facility. All ingredients are Generally Regarded As Safe (GRAS) ingredients. Once produced a full list of allergens and ingredients will be made available. Safety and storage analysis certification will also be available.

1. Animal based protein biscuit containing 12% of total energy as protein (source of protein animal (SA))
2. Plant based protein biscuit containing 12% of total energy as protein (source of protein plant (SP))
3. Animal based protein biscuit containing 20% of total energy as protein (high protein animal (HA))
4. Plant based protein biscuit containing 20% of total energy as protein (high protein plant (HP))
5. A generic taste matched wheat based biscuit (control (C))

Study Outcomes

The products will be assessed for taste, mouth feel and appearance using comparative profiling testing. Data will be recorded using a computerised questionnaire. The questionnaire is internet based so is accessible at multiple sites.

Study design

Each participant will assess each type of product and two control foods twice per session along with one training plate. The layout of the plates will be set as below. Plate order and order of samples on each plate will be advised using a random order as to negate any sequencing bias and samples will be given a randomised number for each plate.

Plate Sample order Training plate SA SP HA HP C Plate 1 SA SP HA HP C Plate 2 SP HA HP C S

Participants

Participants will be recruited from 4 sites, Newcastle University, Bristol University, Aberdeen University and Sheffield University. All participants will be healthy free-living adults. Participants will be recruited to ensure equal gender distribution with groups separated into 40-54, 54-69 and 70+ for analysis. Up to 20 participants of each age group will be required at each site.

ELIGIBILITY:
No allergies to any food Aged over 40

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Taste as assessed by consumer taste panel | Baseline
  Acceptance of taste
Mouth feel as assessed by consumer taste panel | Baseline
  Acceptance of mouth feel
Appearance as assessed by consumer taste panel | Baseline
  Acceptance of mouth feel
Expected satiety as assessed by consumer taste panel | Baseline
  Expected satiety from consuming test biscuits

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - The Rowett Institute, Aberdeen, Aberdeenshire
  - Bristol University, Bristol
  - Department of Oncology & Metabolism, University of Sheffield, Sheffield